CLINICAL TRIAL: NCT02991742
Title: Ioxaglate Versus Iodixanol for the Prevention of Contrast-induced Nephropathy in High-risk Patients After Diagnostic and Therapeutic Cardiac Catheterization (IDPC Trial)
Brief Title: Ioxaglate Versus Iodixanol for the Prevention of Contrast-induced Nephropathy in High-risk Patients (IDPC Trial)
Acronym: IDPC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, RAFAELA ANDRADE PENALVA FREITAS, Principal Investigator, Instituto Dante Pazzanese de Cardiologia
Other Study IDs: 58593116.2.0000.5462
Record Dates: First submitted 2016-12-01; First posted 2016-12-13 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Acute Kidney Failure
Keywords: nephropathy; catheterization; contrast media; ioxaglate; iodixanol; high risk; prevention
MeSH Terms: conditions — Acute Kidney Injury; Kidney Diseases | interventions — Contrast Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Iodixanol: Iodixanol contrast media
  Interventions: Other: contrast media
- Ioxaglate: Ioxaglate contrast media
  Interventions: Other: contrast media

INTERVENTIONS:
Other: contrast media — Compare 2 contrast media
  Other Names: Iodixanol X Ioxaglate

SUMMARY:
Contrast media-induced nephropathy following diagnostic and therapeutic cardiac catheterization.

DETAILED DESCRIPTION:
Contrast-induced acute kidney injury represents a serious complication of procedures requiring administration of iodinated contrast media and is associated with the need for dialysis, prolonged hospitalization, increased costs, and mortality.

Contrast-induced nephropathy is defined as an increase of 25% in serum creatinine before the procedure.

Iodixanol, a nonionic, dimeric, iso-osmolar contrast medium may be less nephrotoxic than low-osmolar contrast media in high-risk patients.

The purpose of this study is to compare iodixanol versus ioxaglate in high risk patients between 48 and 96 hours after procedures that use contrast.

ELIGIBILITY:
Inclusion Criteria:

At least one of the following criteria

* Aged more than 70 years-old
* Chronic renal failure
* Diabetes mellitus
* Congestive heart failure - left ventricular ejection fraction < 0.50
* Shock or intra-aortic ballon pump use
* Urgency or emergency procedures

Exclusion Criteria:

* Patients in dialysis
* Allergy to iodine
* Patient refusal to informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary angiography or percutaneous interventions will be eligible for the trial if they have at least 1 risk factor for contrast-induced acute kidney injury
Sampling Method: Probability Sample
Enrollment: 2262 (Estimated)
Dates: Start 2016-12; Primary Completion 2016-12 (Actual); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Contrast-induced nephropathy incidence | Between 48 and 96 hours after diagnostic and therapeutic cardiac catheterization

SECONDARY OUTCOMES:
Composite of death or need for dialysis in 48 to 96 hours and at 30 days after diagnostic and therapeutic cardiac catheterization | 30 days
  Need for dialysis when patient develop end stage kidney failure -- by the time patient lose about 85 to 90 percent of your kidney function and have a glomerular filtration rate of <15.
The individual components of the combined outcome (total mortality or dialysis indication) | 30 days

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Freitas RAP, Tanajura LF, Mehran R, Chamie D, Chaves A, Centemero M, Braga S, Costa R, Cao D, Sousa A, Feres F, Costa JR Jr. Ioxaglate Versus IoDixanol for the Prevention of Contrast-Induced Nephropathy: The IDPC Trial. J Invasive Cardiol. 2023 Jun;35(6):E281-E290. doi: 10.25270/jic/21.00249. Epub 2023 May 16. PMID 37220640